CLINICAL TRIAL: NCT04884529
Title: Virtual Chair Yoga for Stress in Older Adults (60+) With Mild/Moderate Dementia or Mild Cognitive Impairments and Caregivers (18+) During COVID-19
Brief Title: Virtual Chair Yoga for Older Adults and Caregivers: Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Davis Institute (Other)
Responsible Party: Principal Investigator, Soham Rej MD, MSc, Primary Investigator, Lady Davis Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-2761
Record Dates: First submitted 2021-05-07; First posted 2021-05-13 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Dementia; Mild Cognitive Impairment
Keywords: Dementia; Mild Cognitive Impairments; Caregiving; Stress; Loneliness; Depression; Anxiety; Chair-yoga
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessor will be blinded to participant randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chair Yoga Treatment Group (Experimental): The chair-yoga session will occur for 8-weeks (60 minutes/week) on Zoom. The chair-yoga intervention will include gentle seated postures, relaxation using breathing techniques, and a mindfulness component.
  Interventions: Behavioral: Chair-yoga program
- Waitlist Control Group (No Intervention): These participants will be on a waitlist to receive the chair yoga program after data collection has been completed (e.g., after 8-weeks).

INTERVENTIONS:
Behavioral: Chair-yoga program — 8-week chair yoga program with gentle postures, breathing techniques, and mindfulness.
  Arms: Chair Yoga Treatment Group

SUMMARY:
Over 700,000 Canadians are affected by dementia costing the health care system approximately $10 billion/year. Due to COVID-19, the government has urged individuals over the age of 70 to stay home, putting this population at risk of social isolation. Older adults with mild cognitive impairments (MCIs), dementia, and their caregivers are at an even higher risk of becoming stressed, anxious, and agitated while in lockdown. Unsurprisingly, caregiver burden is extremely common, and often precedes institutionalization of the patient, as the demands of the illness begin to exceed that which the caregiver can sustainably provide. Since social distancing measures have shut down activities and support groups for these individuals, there is an urgent need for scalable, cost-effective, non-pharmacological interventions that can be delivered remotely to improve stress and loneliness. Yoga may be a viable therapeutic modality to address the psychological challenges associated with dementia in patients and caregivers, as it has been shown to decrease stress and improve anxiety and depressive symptoms in various populations. For this reason, the investigators are conducting a randomized controlled trial (RCT) to assess the efficacy of an 8-week virtual chair yoga program to improve stress, psychological symptoms, and caregiver burden. This virtual chair yoga study will engage both older adults with dementia/MCI and caregivers (n=40-60 participants) during COVID-19, which is consistent with the need for decreasing costs and increasing accessibility of novel health interventions during and beyond the pandemic. The investigators will evaluate the effect of this program on stress, loneliness, and mental health related outcomes such as fear of COVID-19, depression, anxiety, and caregiver burden compared to a waitlist control group. There will also be a qualitative component in the form of semi-structured interviews. All quantitative outcomes will be assessed before the program starts and post-intervention and qualitative outcomes will be assessed post-intervention. Participants will be randomly assigned to the treatment group (virtual chair yoga 1 hour per week on Zoom) or the waitlist control group. The investigators hypothesize that after the 8-week yoga program, older adults and caregivers will report lower stress, loneliness, depression, anxiety, fear of COVID-19, and caregiver burden. Results will be available late-2021.

ELIGIBILITY:
Inclusion Criteria for Older Adults:

* Mild cognitive impairment or mild to moderate dementia (MoCA-BLIND score between 8-18 OR a diagnosis from his/her clinician of mild cognitive impairment) or mild to moderate dementia
* Sufficient hearing to follow verbal instructions
* Access to Zoom software and internet connection
* Ability to sit for 60 minutes without discomfort
* At least 60 years old

Exclusion Criteria for Older Adults:

* Severe dementia (MoCA-BLIND score < 8)
* Acute psychotic symptoms
* Acute suicidal ideation or intent
* Resides outside of Quebec

Inclusion Criteria for Caregivers:

* Providing care for someone with cognitive impairments (mild cognitive impairment or mild, moderate, or severe dementia)
* Sufficient hearing to follow verbal instructions
* Access to Zoom software and internet connection
* Ability to sit for 60 minutes without discomfort
* At least 18 years old

Exclusion Criteria for Caregivers:

* Dementia (MoCA-BLIND score < 18)
* Acute psychotic symptoms
* Acute suicidal ideation or intent
* Resides outside of Quebec

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Changes in perceived stress scores as measured by the Perceived Stress Scale (PSS) for treatment group versus control group | Baseline, 8-weeks
  The 8-week randomized controlled trial (RCT) of the virtual chair yoga treatment versus the waitlist control group will assess the effects of the virtual chair yoga on perceived stress in older adults and caregivers, using the PSS.
  Scores on the PSS can range from 0-40, with higher scores indicating higher perceived stress.
  Hypothesis: Following participation in an 8-week RCT of the virtual chair yoga program, older adults with dementia and their caregivers will report lower perceived stress, as measured by the Perceived Stress Scale (PSS) compared to the waitlist control group.

SECONDARY OUTCOMES:
Changes in loneliness scores as measured by the 3-item UCLA Loneliness Scale for treatment group versus control group | Baseline, 8-weeks
  The 8-week randomized controlled trial (RCT) of the virtual chair yoga treatment versus the waitlist control group will assess the effects of the virtual chair yoga on perceived stress in older adults and caregivers, using the PSS.

OTHER OUTCOMES:
Changes in caregiver burden as measured by the Zarit Burden Interview (ZBI) for treatment group versus control group | Baseline, 8-weeks
  The 8-week randomized controlled trial (RCT) of the virtual chair yoga treatment versus the waitlist control group will assess the effects of the virtual chair yoga on caregiver burden in caregivers, using the ZBI.
  Scores on the ZBI can range from 0-88, with higher scores corresponding to higher levels of burden.
  Hypothesis 1: Following participation in an 8-week RCT of the virtual chair yoga program, caregivers of older adults will report less caregiver burden, as measured by the Zarit Burden Interview (ZBI) compared to the waitlist control group.
  Hypothesis 2: Lower scores for older adults on the PHQ-9 and GAD-7 (week 8) will be associated with decreased caregiver burden following participation in an 8-week RCT of the virtual chair yoga program.
Changes in depressive symptoms as measured by the Patient Health Questionnaire-9 (PHQ-9) for treatment group versus control group | Baseline, 8-weeks
  The 8-week randomized controlled trial (RCT) of the virtual chair yoga treatment versus the waitlist control group will assess the effects of the virtual chair yoga on depressive symptoms in older adults and caregivers, using the PHQ-9.
  Scores on the PHQ-9 can range from 0-27, with higher scores indicating more severe depression.
  Hypothesis: Following participation in an 8-week RCT of the virtual chair yoga program, older adults with dementia and their caregivers will report less depressive symptoms, as measured by the Patient Health Questionnaire (PHQ-9) compared to the waitlist control group.
Changes in symptoms of anxiety as measured by the Generalized Anxiety Disorder-7 (GAD-7) scale for treatment group versus control group | Baseline, 8-weeks
  The 8-week randomized controlled trial (RCT) of the virtual chair yoga treatment versus the waitlist control group will assess the effects of the virtual chair yoga on symptoms of anxiety in older adults and caregivers, using the GAD-7.
  Scores on the GAD-7 range from 0-21, with higher scores indicating more severe anxiety.
  Hypothesis: Following participation in an 8-week RCT of the virtual chair yoga program, older adults with dementia and their caregivers will report less symptoms of anxiety, as measured by the Generalized Anxiety Disorder 7-Item Scale (GAD-7) compared to the waitlist control group.
Changes in fear of COVID-19 as measured by the Fear of COVID-19 scale (FC-19S) for treatment group versus control group | Baseline, 8-weeks
  The 8-week randomized controlled trial (RCT) of the virtual chair yoga treatment versus the waitlist control group will assess the effects of the virtual chair yoga on fear of COVID-19 in older adults and caregivers, using the FC-19S.
  Scores on the FC-19S range from 7-35, with higher scores indicating more fear of COVID-19.
  Hypothesis: Following participation in an 8-week RCT of the virtual chair yoga program, older adults with dementia and their caregivers will report less fear of COVID-19, as measured by the Fear of COVID-19 scale (FC-19S) compared to the waitlist control group.
Semi-structured interviews/focus groups for the Qualitative Component | 8-weeks
  The 8-week randomized controlled trial (RCT) of the virtual chair yoga treatment versus the waitlist control group will assess lived experiences and perceptions from baseline to 8-weeks in the form of interview/focus groups.
Changes in mindfulness as measured by the 5 Facet Mindfulness Questionnaire: Short form (FFMQ-SF) for treatment group versus control group. | Baseline, 8-weeks
  The 8-week randomized controlled trial (RCT) of the virtual chair yoga treatment versus the waitlist control group will assess the effects of the virtual chair yoga on levels of mindfulness in older adults and caregivers, using the FFMQ-SF.
  Scores on the FFMQ-SF range from 0-120, with higher scores indicating higher levels of mindfulness.
  Hypothesis: Following participation in an 8-week RCT of the virtual chair yoga program, older adults with dementia and their caregivers will report higher levels of mindfulness, as measured by the 5 Facet Mindfulness Questionnaire: Short form (FFMQ-SF) compared to the waitlist control group.
Changes in levels of self-compassion as measured by the Self-Compassion Scale-Short Form (SCS-SF) for treatment group versus control group. | Baseline, 8-weeks
  The 8-week randomized controlled trial (RCT) of the virtual chair yoga treatment versus the waitlist control group will assess the effects of the virtual chair yoga on levels of self-compassion in older adults and caregivers, using the SCS-SF.
  Scores on the SCS-SF range from 0-60, with higher scores indicating higher levels of self-compassion.
  Hypothesis: Following participation in an 8-week RCT of the virtual chair yoga program, older adults with dementia and their caregivers will report higher levels self-compassion, as measured by the Self-Compassion Scale-Short Form (SCS-SF) compared to the waitlist control group.
Changes in levels of rejection sensitivity as measured by the Rejection Sensitivity Questionnaire - Adult Version (A-RSQ) for treatment group versus control group. | Baseline, 8-weeks
  The 8-week randomized controlled trial (RCT) of the virtual chair yoga treatment versus the waitlist control group will assess the effects of the virtual chair yoga on rejection sensitivity in older adults and caregivers, using the A-RSQ.
  Hypothesis: Following participation in an 8-week RCT of the virtual chair yoga program, older adults with dementia and their caregivers will report less sensitivity to rejection, as measured by the Rejection Sensitivity Questionnaire - Adult Version (A-RSQ) compared to the waitlist control group.
Changes in levels of social pleasure and positive emotions as measured by the Social Safeness and Pleasure Scale (SSPS) for treatment group versus control group. | Baseline, 8-weeks
  The 8-week randomized controlled trial (RCT) of the virtual chair yoga treatment versus the waitlist control group will assess the effects of the virtual chair yoga on levels of social pleasure and positive emotions in older adults and caregivers, using the SSPS.
  Hypothesis: Following participation in an 8-week RCT of the virtual chair yoga program, older adults with dementia and their caregivers will report higher levels of social pleasure and positive emotions, as measured by the Social Safeness and Pleasure Scale (SSPS) compared to the waitlist control group.
Changes in perceptions of social connectedness as measured by the Social Connectedness Scale-Revised (SCS) for treatment group versus control group. | Baseline, 8-weeks
  The 8-week randomized controlled trial (RCT) of the virtual chair yoga treatment versus the waitlist control group will assess the effects of the virtual chair yoga on perceptions of social connectedness in the individuals social environment for older adults and caregivers, using the SCS.
  Hypothesis: Following participation in an 8-week RCT of the virtual chair yoga program, older adults with dementia and their caregivers will report higher perceptions of social connectedness in their environment, as measured by the Social Connectedness Scale-Revised (SCS) compared to the waitlist control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Community and Family Psychiatry, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No